CLINICAL TRIAL: NCT02192060
Title: Efficacy of a Triclosan Formulation to Control the Initial Subgingival Biofilm Formation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Rui Vicente Oppermann, DDS, PhD, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: RVOppermann01
Record Dates: First submitted 2013-11-13; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Dental Plaque
Keywords: Biofilm; Triclosan; Crossover; Clinical trial
MeSH Terms: conditions — Dental Plaque | interventions — Triclosan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Using of a suspension containing Triclosan
  Interventions: Other: Test - Using of a suspension containing Triclosan
- Control (Placebo Comparator): Using of a suspension without Triclosan or other active ingredient
  Interventions: Other: Control - Using of a suspension without Triclosan

INTERVENTIONS:
Other: Test - Using of a suspension containing Triclosan — The participants should have used only the suspension containing Triclosan during 5 days and have stopped with their biofilm control homemade procedures.
  Arms: Test
Other: Control - Using of a suspension without Triclosan — The participants should have used only the Placebo suspension during 5 days and have stopped with their biofilm control homemade procedures.
  Arms: Control

SUMMARY:
The aim of the study is to compare the effect of a suspension containing Triclosan in dynamic of the subgingival biofilm formation versus a Placebo suspension. The initial subgingival biofilm formation will be evaluated by means of Plaque Free Zone (PFZ).

DETAILED DESCRIPTION:
This is a double blind, cross over, randomized clinical trial. 28 volunteers will stop mechanical supragingiva biofilm removal measures for 96h following a complete scaling and polishing of the tooth surfaces. During this period they will be asked to rinse for one minute with a slurry of either a triclosan containing dentifice or a control without triclosan. Every 24h the presence of deposits will be registered with special atention to the presence of a plaque free zone between the apical border of the deposits and the gingival margin. Absence of deposits is scored 0, presence of deposits and plaque free zone =1 and presence of deposits and absence of plaque free zone =2 (MALISKA, A. N. et al. Measuring early plaque formation clinically. Oral health preventive dentistry, v. 4, p. 273-278, 2006). The prevalence of scores and the rate of changes from scores 0 and 1 into 2 will be evaluated for significance. Sample size was calculated taking the results from the study o MALISKA, AN (2006) as reference.

ELIGIBILITY:
Inclusion Criteria:

* age from 18 years;
* non-smokers;
* have good general health;
* present at least 20 natural teeth in the mouth, including the incisors, canines and premolars without restorations, crowns, gingival recession, anatomic defects, gingivitis e/or periodontitis.

Exclusion Criteria:

* positive history of using antibiotic e/or anti-inflammatory drugs in the month previous to the initial consultation;
* positive history of allergies at using Triclosan;
* pregnant or lactating patients;
* patients in use of fixed orthodontic appliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Presence of Plaque Free Zone | 24 hours
  The presence of scores 0, 1 or 2 of the index "Plaque Free Zone" will be recorded at baseline and at each 24 hours, during a period of 96 hours (4 days).

CONTACTS AND LOCATIONS:
Overall Officials: Rui V. Oppermann, DDS, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Dentistry Faculty, Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil